CLINICAL TRIAL: NCT03206853
Title: Clinical Trail of Hybrid Operating Technique in Management of Complex Intracranial Aneurysms With Coexistence of Multiple Risk Factors
Brief Title: Surgical Management of Complex Intracranial Aneurysms With Hybrid Operating Techniques
Acronym: CIA-HOTs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: liuxingju (Other Government)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Sponsor-Investigator, liuxingju, Researcher, Ministry of Science and Technology of the People´s Republic of China
Organization: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BJTTH-004
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Intervention Model Description: Traditional therapy group：the aneurysms will be executed by traditional procedure, including microsurgical clipping, endovascular coiling or stenting, etc.
  Hybrid operation group: Intervene with hybrid operating techniques, eg. microsurgical clipping+endovascular coiling or with the assistant of balloon occlusion.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid operation group (Experimental): Intervene with hybrid operating techniques, eg. microsurgical clipping+endovascular coiling or with the assistant of balloon occlusion.
  Interventions: Procedure: Hybrid Operating Techniques
- Traditional therapy group (Other): The aneurysms will be executed by traditional procedure, including microsurgical clipping, endovascular coiling or stenting, etc.
  Interventions: Procedure: Hybrid Operating Techniques

INTERVENTIONS:
Procedure: Hybrid Operating Techniques — It is a cooperation of existing endovascular interventional techniques and microsurgical techniques. Different from traditional management, hybrid operating techniques make it possible for 2 existing techniques conducting simultaneously in a hybrid operating theater. It optimizes the traditional microsurgical techniques for complex intracranial aneurysms and avoids the transportation of patients and the risks of intervals between stages in traditional ones. It includes balloon-assisted parental arterial occlusion, one-stage aneurysm clipping/wrapping/isolation and embolization/diverter implantation, etc.
  Other Names: microsurgical clipping; microsurgical dissection; microsurgical wrapping; microsurgical isolation; endovascular coiling; balloon-assisted occlusion; flow diverter

SUMMARY:
To evaluate the clinical benefits and risks of hybrid operating techniques in management of complex intracranial aneurysms, which could coexists with multiple risk factors.

DETAILED DESCRIPTION:
Purpose: Have an evaluation of clinical benefits and risks of hybrid operating techniques in management of complex intracranial aneurysms (CIAs), which could coexists with multiple risk factors. Meanwhile, as a new cooperative interventional modality, optimized workflows, technical key knots and operation routines will be explored in the study.

Objects: Patients with CIAs, coincident with inclusion and exclusion criterion and admitted in participating organizations.

Methods: Patients will be distributed into 2 groups, including traditional therapy group(control group) and hybrid operating group(trial group), and conduct with traditional neurosurgical management or one-stage hybrid operating management correspondingly. Peri-operative mortality rate is considered to be the primary observing indicator, and morbidity rate of peri-operative cerebral hemorrhagic/ischemic event, morbidity rate of aneurysmal residuals, morbidity rate of neural functional deteriorations, and health-economic indicators are secondary indicators.The information of operations will be recorded in detail as evidence of optimization of workflow and technical key knots.

ELIGIBILITY:
Inclusion Criteria:

* with diagnosed complex intracranial aneurysm by digital subtraction angiography(DSA);
* got SAH in history;
* neural functional deficits due to aneurysms;
* with <4 in Hunt-Hess Grades;
* ≥5.0mm in the maximum diameter;
* <70 years old;
* with irregular morphological features and high rupture risk.

Exclusion Criteria:

* >70 in age, with low rupture risk;
* cannot tolerant the operation;
* patient or relative refuses to participate the trail;
* SAH patient with ≥4 Hunt-Hess grading system;
* <5.0mm in the maximum diameter.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
operation-related mortality rate | From the time of operation begin to 48 hours after operation
  the mortality rate related to the operation

SECONDARY OUTCOMES:
Morbidity rate of peri-operative intracranial hemorrhage | From date of admission to the 7 days after operation
  Intracranial hemorrhagic events happening during the peri-operative period, including subarachnoid hemorrhage, intracranial hemorrhage, intraventricular hemorrhage caused by the rupture of aneurysms with neuro-imaging evidence.
Morbidity rate of peri-operative intracranial ischemic events | From date of admission to 7 days after operation
  The intracranial ischemic events happening during the peri-operative period, including operation-related infarction, embolization, etc. With neuro-imaging evidence.
Residual rate of aneurysms | the date of first post-operative cerebrovascular angiography is conducted, up to 3 months after operation
  the morbidity rate of aneurysmal residue, with post-operative DSA/CTA evidence
Morbidity rate of neural functional deterioration in 48 hours after operation | 48 hours after operation, ±6 hours
  The score of modified Rankin Scale increases ≥2, comparing to the original mRS scores
Morbidity rate of neural functional deterioration in 7 days | 7 days after operation, ±2 days
  The score of modified Rankin Scale increases ≥2, comparing to the original mRS scores
Morbidity rate of neural functional deterioration in 3 months | the 3rd month after operation, ±1 week
  The score of modified Rankin Scale increases ≥2, comparing to the original mRS scores
Morbidity rate of neural functional deterioration in 6 months | the 6th month after operation, ±1 week
  The score of modified Rankin Scale increases ≥2, comparing to the original mRS scores
Morbidity rate of neural functional deterioration in 12 months | the 12th month after operation, ±1 week
  The score of modified Rankin Scale increases ≥2, comparing to the original mRS scores
Treatment-related costs | through study completion, an average of 1 year
  All expenses cost in hospital relating to the aiming disease
Duration of hospitalization | through study completion, an average of 1 year
  Total hospitalization of all stages of treatments to IAs, including admissions for evaluation, operation, and DSA
Duration of total operating time | through study completion, an average of 1 year
  Total operating time of all procedures, including operation, and DSA

CONTACTS AND LOCATIONS:
Overall Officials: Jizong Zhao, MD, Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
the IPD will be open to public researchers in 6 months after the study closed.